CLINICAL TRIAL: NCT02038686
Title: Treatment of Unstable 31.A2 and 31.A3 Trochanteric Fractures. Randomised Comparison of the Proximal Femoral Nail PFN-A Short and the PFN-A Long.
Acronym: PFN-A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ferran Fillat Gomà (Other)
Collaborators: Parc Taulí Hospital Universitari (Other)
Responsible Party: Sponsor-Investigator, Ferran Fillat Gomà, Medical Doctor, Corporacion Parc Tauli
Organization: Corporacion Parc Tauli (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPTCOT2013/01
Record Dates: First submitted 2014-01-15; First posted 2014-01-16 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Unstable Proximal Femoral Fracture
Keywords: Hip fracture; Unstable (31A2 and 31A3); Proximal femoral nail
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard PFN-A (Active Comparator): Patients with unstable proximal femoral fractures treated with PFN-A short nail (170-240mm)
  Interventions: Device: PFN-A
- Long PFN-A (Active Comparator): Patients with unstable proximal femoral fractures treated with PFN-A long nail (300-420mm)
  Interventions: Device: PFN-A

INTERVENTIONS:
Device: PFN-A
  Other Names: Proximal femoral nail Synthes

SUMMARY:
1. Introduction:

   Controversy exists with regard to whether to treat AO/OTA (Orthopaedic Trauma Association) 32.A2 - 32-A3 fractures of the proximal part of the femur with an intramedullary short PFN-A or long PFN-A. A prospective, randomized, controlled trial is performed to compare the outcome treatment of these unstable fractures of the proximal part of the femur with either a short PFN-A (170-240mm) or long PFN-A (300-420mm).
2. Objectives and Hypothesis The hypothesis is that the Short PFN-A would have fewer complications than Long PFN-A

   Main Objective: Is defined as Total number of complications between PFN-A short and PFN-A long. Outcome measures were subdivided into preoperative, perioperative and post-operative. Follow up data at four weeks, three months and one year.

   Secondary objectives: Complete and uneventful radiological and clinical healing of the fracture. Revision operations (related to the failure of primary treatment) and mortality. Baseline characteristics were documented pre-operatively: Outcome measures were subdivided into intra-operative, post-operative and follow up data at four weeks, three months and one year.
3. Methodology: One hundred and eighty eight patients presenting with an AO/OTA 31-A2 and 31-A3 fracture of the proximal part of the femur will be randomized, at the time of the admission, to fixation with use either a short PFN-A or a long PFN-A.

ELIGIBILITY:
Inclusion Criteria:

* Patients 60 years old above.
* Patients with trochanteric fracture 31.A2 and 31.A3 AO classification for long bones
* Patients that accept to participate on the study under consent

Exclusion Criteria:

* Metaphyseal fractures with extension more than 3 cm in reference to lesser trochanter calibrated and analyzed with PreOPlan registered application.
* Combination of fractures in the proximal femur.
* Pathological fractures.
* Diaphyseal femoral fractures.
* Rejection of surgery by the patient.
* Contraindications to the use of either implants studied.
* Patients who do not wish to participate in this study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Total number of complications between PFN-A short and PFN-A long | One year
  follow-up data is recruited at 4 weeks, 3 months and one

SECONDARY OUTCOMES:
Complete and uneventful radiological and clinical healing of the fracture and mortality | One year
  follow-up data is recruited at 4 weeks, 3 months and one year.

CONTACTS AND LOCATIONS:
Overall Officials: Ferran Fillat-Gomà, MD, Principal Investigator — Hospital Universitario Parc Tauli de Sabadell; Joan Murias-Álvarez, MD, Study Director — Hospital Universitario Parc Tauli de Sabadell
Locations (1):
- Hospital Universitario Parc Taulí de Sabadell, Sabadell, Barcelona, Spain